CLINICAL TRIAL: NCT06143631
Title: Letrozole for Treatment of Uterine Fibroids: A Randomized, Placebo-Controlled Trial
Brief Title: Prescription of Letrozole for Uterine Myoma
Acronym: PLUM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-39255; R01HD112465 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Leiomyoma, Uterine; Leiomyoma; Fibroid; Fibroid Uterus
MeSH Terms: conditions — Leiomyoma | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): Oral letrozole 2.5mg/day
  Interventions: Drug: Letrozole 2.5mg
- Placebo and Letrozole (Placebo Comparator): Placebo capsule for 12 weeks; Oral letrozole 2.5mg/day for 12 weeks
  Interventions: Drug: Letrozole 2.5mg; Other: Placebo

INTERVENTIONS:
Drug: Letrozole 2.5mg — Oral letrozole 2.5mg/day
Other: Placebo — Placebo capsule
  Arms: Placebo and Letrozole

SUMMARY:
The PLUM Study is a randomized, double-blinded, 2-arm, parallel-group, placebo-controlled trial is designed to compare the efficacy of letrozole versus placebo on leiomyoma-related symptoms and quality of life as well as leiomyoma and uterine size.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 and less than 54 years of age (to focus on an adult, premenopausal population)
* Female sex, based on sex identified on their birth certificate (no other gender requirements)
* Have uterine leiomyomata that have been visualized on pelvic imaging (i.e., ultrasound or MRI) in the last 24 months
* Report symptoms associated with leiomyomata such as heavy uterine bleeding, pelvic pressure or discomfort, urinary or bowel abnormalities, or dyspareunia for the past 3 months
* Have at least moderate leiomyomata symptom burden, with UFS-QOL SSS score of 30 or higher at baseline
* Has regularly occurring menstrual periods of ≤ 14 days duration with a cycle of 21 to 38 days from the start of one menstrual period until the start of the next, by patient history for at least 3 months prior to screening
* Agree to use a non-hormonal or barrier method of contraception with any sexual activity with a non-sterile male partner during the study period (i.e., use of copper IUD is consistent with eligibility)

Exclusion Criteria:

* Screening pelvic imaging indicating any leiomyomata ≥10 cm in maximum diameter, or uterine size ≥16 cm in length (equivalent to 16 weeks gestation)-note that candidates who exclusively have prior clinical pelvic imaging 12-24 months ago will be excluded if imaging includes leiomyomata ≥9 cm in maximum diameter, or uterine size ≥15 cm in length, presuming leiomyoma growth of ≥1 cm per year
* Screening pelvic imaging indicating only one, sole leiomyoma <2 cm in maximum diameter
* Any submucosal leiomyoma that is >50% within uterine cavity (FIGO Type 0 or Type 1 leiomyomata)
* Visit to the emergency room or hospitalization for leiomyoma symptoms in the last 12 weeks
* Leiomyomata treated by surgery, radiologic procedure in the last 12 weeks; or plans to undergo any of the above in the next 24 weeks
* Leiomyomata treated by GRNH agonist or antagonist in the last 12 weeks; or plans to use the above in the next 24 weeks
* Currently pregnant or lactating, pregnant or lactating in the past 12 weeks, or planning to become pregnant in the next 24 weeks
* Screening serum hemoglobin <8 g/dL, or history of blood transfusion in the last 12 weeks (indicating severe anemia)
* Screening cholesterol lipid panel testing showing LDL cholesterol level ≥ 190 mg/dL (due to rare side effects over long-term use of aromatase inhibitors in postmenopausal women)
* Screening serum estradiol level <30 pg/mL (consistent with postmenopausal status)
* Irregularly timed bleeding, including bleeding or spotting in between periods, in the past 3 months.
* History of osteoporosis (based on self-reported DEXA indicating bone mineral density Z-score < -2.0 at spine, total hip, or femoral neck; a prior fracture judged to be a fragility fracture; or self-reported use of bisphosphonates, calcitonin, calcitriol, ipriflavone, teriparatide, or denosumab for bone density loss)
* History of severe liver disease (Child Pugh Class C cirrhosis), posing safety risks for use of letrozole
* Current or prior history of breast cancer (given potential need to take letrozole for breast cancer treatment or secondary prevention)
* Screening pelvic imaging indicating an Ovarian-Adnexal Reporting and Data System (O-RADS) category 3, 4, or 5 ovarian or adnexal lesion
* Screening pelvic imaging concerning for other current cancer of the gynecologic, genitourinary or gastrointestinal system
* Prior hypersensitivity or significant adverse reaction to letrozole or any aromatase inhibitor, or to an ingredient in the placebo capsule
* Use of letrozole, other aromatase inhibitor, or selective estrogen receptor modulator (SERM) medications in the past 4 weeks, or existing plans to initiate one of these in the next 24 weeks
* Use of oral, vaginal, or topical exogenous estrogen, progestin, or androgen therapy in the past 4 weeks; or injectable forms of the above in the past 12 weeks; or plans to initiate any of the above in the next 24 weeks
* Use of medications with potential unsafe interactions with letrozole in the past 4 weeks (methadone, levomethadone, nintedanib, thalidomide), or plans to initiate these in the next 24 weeks
* Any condition that, in the opinion of the investigators, would interfere with ability to complete study procedures, including acute or uncontrolled mental health condition, substance abuse, or inability to complete procedures in English (or Spanish, for sites that offer study assessments in Spanish)

Ages: 21 Years to 53 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Uterine leiomyoma-related symptom severity over 12 weeks of treatment | Baseline to 12 weeks
  Change in Uterine Fibroid Symptoms Quality of Life (UFS-QOL) Symptom Severity Scale (SSS) score [Range 8-40 with higher score indicating worse symptoms and worse outcomes]

SECONDARY OUTCOMES:
Uterine leiomyoma-related quality of life over 12 weeks of treatment | Baseline to 12 weeks
  Change in Uterine Fibroid Symptoms Quality of Life (UFS-QOL) Health-Related QOL component score [Range 29-145 points, with higher score indicating better QoL and better outcomes]
Total leiomyoma volume over 12 weeks of treatment | Baseline to 12 weeks
  Change in total leiomyoma volume based on pelvic ultrasound measurements
Total uterine volume over 12 weeks of treatment | Baseline to 12 weeks
  Change in total uterine volume based on pelvic ultrasound measurements
Symptoms of heavy menstrual bleeding | Baseline to 12 weeks
  Change in symptoms of heavy menstrual bleeding based on a modified Menstrual Bleeding Questionnaire (MBQ) score [Range 0-48 with higher MBQ score indicating worse symptoms and a negative impact on quality of life]
Improvement in Sexual Functioning | Baseline to 12 weeks
  Change in pelvic problems-related sexual function as measured by the Sexual Health Outcomes in Women Questionnaire (SHOW-Q) Pelvic Problems Interference subscale score [Range 0-100 with higher scores indicating better sexual function]
Symptoms of pelvic pain | Baseline to 12 weeks
  Change in pelvic pain severity/intensity "on average" (evaluated on a standard numerical rating scale of 0-10, lower rating indicating better outcomes and less pain)
Symptoms of urogenital distress | Baseline to 12 weeks
  Change in distressing urogenital symptoms such as urinary frequency, urinary incontinence, and genital pain, as measured by Urogenital Distress Inventory-6 (UDI-6) [Range 0-100 with higher scores indicating higher disability/worse outcomes]
Effect of letrozole on serum cholesterol levels | Baseline to 12 weeks
  Change in serum LDL cholesterol levels
Effect of letrozole on serum estradiol levels | Baseline to 12 weeks
  Change in serum estradiol levels
Effect of letrozole on frequency of hot flashes | Baseline to 12 weeks
  Change in frequency of vasomotor symptoms (hot flashes) as measured by the Hot Flush Rating Scale (HFRS) [no scale range but less # of reported hot flashes indicates better outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, MAS, Principal Investigator — University of California, San Francisco; Alison Huang, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No